CLINICAL TRIAL: NCT04180098
Title: Improving Gait Adaptability in Hereditary Spastic Paraplegia During Task-specific Training on the C-Mill: Towards Evidence-Based and Individually Tailored Rehabilitation
Brief Title: Improving Gait Adaptability in Hereditary Spastic Paraplegia
Acronym: Move-HSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Jacques and Gloria Gossweiler Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 108836
Record Dates: First submitted 2019-11-20; First posted 2019-11-27 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-03

CONDITIONS: Hereditary Spastic Paraplegia; Strumpell Disease
Keywords: hereditary spastic paraplegia; C-mill; gait adaptability; rehabilitation
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Spastic paraplegia 3, autosomal dominant

STUDY DESIGN:
Intervention Model Description: All participants monitor their physical activity for 1 week, and falls for 15 weeks. After the screening, participants are randomized. Gait and balance capacity will be assessed in the movement lab of Radboudumc. Participants in the intervention group receives 5 weeks of C-mill training, which is immediately followed by an assessment in the movement lab, one-week of activity monitoring and fall monitoring during a 15 week follow-up period. After follow-up they will receive a final assessment in our movement lab. Participants in the control (waiting list) intervention, continue usual care for 5 weeks, followed by an assessment in the movement lab and one-week of activity monitoring. Subsequently, they receive 5 weeks of C-mill training, followed by an assessment in the movement lab, one-week of activity monitoring and fall monitoring in a follow-up period of 15 weeks. After follow-up, they receive a final assessment in the movement lab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Context specific C-mill training (Experimental): Five week C-mill training on gait adaptability.
  Interventions: Behavioral: C-mill intervention
- Usual care (Other): Usual care for participants with HSP. May vary per individual.
  Interventions: Behavioral: C-mill intervention; Other: No intervention

INTERVENTIONS:
Behavioral: C-mill intervention — A five week personalised rehabilitation program. Participants train gait adaptability via obstacle negotiation, precision stepping and unexpected accelerations and decelerations. The strategies are trained in a safe environment on the C-mill, a treadmill providing augmented reality via visual and acoustic cues. The treatment is implemented in a five week period via 10 biweekly sessions. Each treatment session lasts 60 minutes. In total, participants will receive C-mill training for a total of ten hours. The training will be carried out by a skilled physiotherapist.
Other: No intervention — Participants in the control group are placed on a waiting list.
  Arms: Usual care

SUMMARY:
This study evaluates the effects of ten hours C-mill training on gait adaptability in participants with hereditary spastic paraplegia (HSP). Half of the participants start with five weeks of C-mill training (ten 1-hour sessions). The other participants are placed on a waiting list, which is followed by the same five weeks of C-mill training (ten 1-hour sessions). It is hypothesized that ten hours of context specific C-mill training is effective in improving gait adaptability in participants with pure HSP.

DETAILED DESCRIPTION:
Hereditary spastic paraplegia (HSP) is a relatively common, slowly progressive movement disorder that seriously impacts on gait capacity. Patients with HSP experience incremental muscle stiffness, muscle weakness and balance problems and, as a consequence, increasing difficulties to adjust their gait pattern to changing environmental demands. This is a major problem as such 'gait adaptability' is critical for independent and safe mobility in daily life. Impaired gait adaptability will also result in falls and fall-related injuries and reduce quality of life. Therefore, there is an urgent need for evidence-based rehabilitation interventions to improve gait adaptability in patients with HSP. Participants train gait adaptability via obstacle negotiation, precision stepping and unexpected accelerations and decelerations. The strategies are trained in a safe environment on the C-Mill, a treadmill providing augmented reality via visual and acoustic cues.

Objectives

This study aims to promote an essential step towards evidence-based and individually tailored gait rehabilitation in participants with hereditary spastic paraparesis. The objectives are twofold:

1. To study the effect of ten 1-hour sessions C-Mill training on gait adaptability in participants with pure-HSP.
2. To study the effect of ten 1-hour sessions C-Mill training on spatiotemporal and functional capacity parameters and to identify key-determinants of C-Mill training efficacy in participants with pure-HSP.

It is hypothesized that ten hours of context specific C-mill training is effective in improving gait adaptability in participants with pure HSP, as measured with the obstacle subtask of the emory functional ambulation profile (E-FAP).

Sample size calculation is based on previous studies concerning the effects of gait adaptability interventions on the obstacle subtask of the E-FAP. A total of 32 participants is sufficient to demonstrate an expected improvement on the obstacle subtask score of the E-FAP. To allow a 10% attrition rate, 36 participants will be included.

Participants will be recruited from the Radboud Expert Centre of Genetic Movement Disorders (part of the ERN-RND) which has specific HSP expertise. The treating physician of the patient will ask whether the investigator may contact the patient. Furthermore, mailings through the HSP patient group, that is part of the patient organization "Spierziekten Nederland", will be sent to their members with HSP. If patients are interested in participating, they can contact the investigator and will be informed via an information letter (to which the informed consent form is attached). Participants will then have two weeks to consider their decision whether to participate. After the two week period, the investigator will contact them about their decision.

Data will be coded numerically (e.g. HSP01, HSP02) and an identification code list will be used to link the data to the participant. The key to the code will be safeguarded by the investigators. The project leader and all other investigators will have access to the source data. Data will be kept for fifteen years. The handling of data will comply with the Dutch Personal Data Protection Act and participants' privacy will be protected. The monitoring will be performed according to NFU guidelines for negligible risk intensity.

Descriptive data analysis will be used to outline characteristics of both intervention groups. The effect of gait adaptability training on primary and secondary outcomes will be tested using ANCOVA. Post-intervention measurements will be used as dependent variables and Group (C-Mill versus waiting list) and pre-intervention measurements as independent between-subjects factors. Time will be tested as a within-subjects factor. The retention of gait adaptability training will be tested by merging both groups and using a repeated measures ANOVA with Time as a within-subjects factor (C-Mill group: measurements 1, 2 and 3; waiting list: measurements 2, 3 and 4). Post-hoc tests will be performed in the case of significant main or interaction effects, using paired t-tests. Fall rates will be processed descriptively. Depending on the distribution of the data, the rate of near falls may be analyzed using Wilcoxon signed rank test. In addition, to determine key determinants of C-Mill training efficacy, a stepwise linear regression analysis will be performed with training-induced change in gait adaptability (relative change of the obstacle subtask of the E-FAP) as the dependent variable. Univariate analyses will be performed to select the best factors from the available demographic and clinical characteristics.

Adverse events All adverse events reported spontaneously by the participants or observed by the investigator or his staff will be recorded. The sponsor will report the SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within seven days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of 8 days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after the sponsor has first knowledge of the serious adverse events. The risk associated with participation will be negligible, according to the risk classification of the NFU. Burden associated with the measurements will be limited, as the number of measurements will be relatively low.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of pure-HSP based on molecular diagnosis or based on inheritance pattern
* Aged between 18-70 years old
* Being able to walk barefoot on a level ground for 50 meters without a walking aid (use of orthopaedic devices or made-to-measure footwear is allowed).

Exclusion criteria:

* Other neurological or serious orthopaedic or psychiatric co-morbidity
* Previous HSP-related surgical interventions of the lower extremities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
The mean changes in time scores of the obstacle subtask of the emory functional ambulation profile | Pre-intervention (week 0) till post-intervention (week 6)
  Patients are asked to negotiate a ten meter obstacle course. The number of seconds it takes to complete the subtask is recorded, and multiplied by a factor corresponding to the level of assistive devices used. A lower time score indicates better obstacle negotiation

SECONDARY OUTCOMES:
The mean change in the time score on the ten meter walk test | Pre-intervention (week 0) till post-intervention (week 6)
  The ten meter walk test (10MWT) is a standardised and recommended measurement of walking velocity. Patients walk ten meters in a straight line: three times at a comfortable speed, and three times as fast as possible, whilst keeping safety in mind. The number of seconds it takes to walk ten meters is recorded.
The mean change of the mini balance evaluation system | Pre-intervention (week 0) till post-intervention (week 6)
  The mini balance evaluation system (mini-BEST) is a 14-item, 3 points ordinal rating scale (0-2 points) to evaluate balance performance in 4 subcategories: anticipatory postural control, reactive postural control, sensory orientation and stability in gait. The attainable scores ranges from 0-28 points, in which a higher score indicates a higher balance performance.
Mean changes of activity levels measured as time spent active of passive during 24 hours | Pre-intervention (week 0) till post-intervention (week 6)
  Physical activity levels of daily life will be registered via the Activ8 Monitor. The monitor consists of 3 axial accelerometers that is worn on the upper thigh. It registers body positions (lying/non-wear/sitting and standing) and activities (walking, running, cycling).
The mean changes in scores of the activities specific balance confidence scale | Pre-intervention (week 0) till post-intervention (week 6)
  Balance confidence will be measured via the activities-specific balance confidence scale. This subjective questionnaire consisting of sixteen indoor and outdoor situations. Patients are asked to express their confidence to safely execute to proposed situations without falling. Scores range from 0-100 in which a higher scores indicates more confidence.
Mean changes in number of falls and near falls | Pre-intervention (week 0) and after the follow-up period of fifteen weeks (experimental group week 21, control group week 27)
  Patients are asked to monitor their falls and near falls via a fall calendar. Patients are asked to fill in when the (near) fall occurred, a short description of the event and if the patients was injured.
The mean change in the time score on the walking adaptability ladder test | Pre-intervention (week 0) till post-intervention (week 6)
  The walking adaptability ladder test (WALT) is a novel test for measuring stepping precision. A standardised ladder is placed on the floor. It consists of 19 rectangular planes which gradually decrease two centimetres in length (range: 64cm - 28cm). Patients starts in the biggest plane and walk as fast as possible to the other side, turn and return to the biggest plane whilst avoiding the ladder rungs. Scoring is via a time score: faster is indicative of better stepping precision. Patients perform the test four times: Twice with one feet per plane, and twice with both feet in one plane.
Mean changes in spatio-temporal gait parameters | Pre-intervention (week 0) till post-intervention (week 6)
  Gait analysis is performed at the movement lab (Radboudumc, Nijmegen). Spatio-temporal parameters are assessed during a 3D full body gait analysis using the VICON analysis system ((©Vicon Motion Systems Ltd., London, UK). Eight infrared cameras measured the coordinates of the reflective markers. The following temporal gait parameters are assessed: stride length (m), step length (m), step width (m), duration of swing time (%), stance time (%), single support (%) and double support (%). Participants walk at their self-selected and maximum speed over a 10 meter walkway. A total of 3 trials per condition is recorded.

OTHER OUTCOMES:
The mean changes in time scores of the obstacle subtask of the emory functional ambulation profile | Pre C-mill intervention (experimental group week 0, control group week 6), post C-Mill intervention (experimental group week 6, control group week 12) and after the follow-up period of fifteen weeks (experimental group week 21, control group week 27)
  Patients are asked to negotiate a ten meter obstacle course. The number of seconds it takes to complete the subtask is recorded, and multiplied by a factor corresponding to the level of assistive devices used. A lower time score indicates better obstacle negotiation
The mean change in the time score on the ten meter walk test | Pre C-mill intervention (experimental group week 0, control group week 6), post C-Mill intervention (experimental group week 6, control group week 12) and after the follow-up period of fifteen weeks (experimental group week 21, control group week 27)
  The ten meter walk test (10MWT) is a standardised and recommended measurement of walking velocity. Patients walk ten meters in a straight line: three times at a comfortable speed, and three times as fast as possible, whilst keeping safety in mind. The number of seconds it takes to walk ten meters is recorded.
The mean change of the mini balance evaluation system | Pre C-mill intervention (experimental group week 0, control group week 6), post C-Mill intervention (experimental group week 6, control group week 12) and after the follow-up period of fifteen weeks (experimental group week 21, control group week 27)
  The mini balance evaluation system (mini-BEST) is a 14-item, 3 points ordinal rating scale (0-2 points) to evaluate balance performance in 4 subcategories: anticipatory postural control, reactive postural control, sensory orientation and stability in gait. The attainable scores ranges from 0-28 points, in which a higher score indicates a higher balance performance.
Mean changes of activity levels measured as time spent active of passive during 24 hours | Pre C-mill intervention (experimental group week 0, control group week 6) and post C-Mill intervention (experimental group week 6, control group week 12)
  Physical activity levels of daily life will be registered via the Activ8 Monitor. The monitor consists of 3 axial accelerometers that is worn on the upper thigh. It registers body positions (lying/non-wear/sitting and standing) and activities (walking, running, cycling).
The mean changes in scores of the activities specific balance confidence scale | Pre C-mill intervention (experimental group week 0, control group week 6), post C-Mill intervention (experimental group week 6, control group week 12) and after the follow-up period of fifteen weeks (experimental group week 21, control group week 27)
  Balance confidence will be measured via the activities-specific balance confidence scale. This subjective questionnaire consisting of sixteen indoor and outdoor situations. Patients are asked to express their confidence to safely execute to proposed situations without falling. Scores range from 0-100 in which a higher scores indicates more confidence.
The mean change in the time score on the walking adaptability ladder test | Pre C-mill intervention (experimental group week 0, control group week 6), post C-Mill intervention (experimental group week 6, control group week 12) and after the follow-up period of fifteen weeks (experimental group week 21, control group week 27)
  The walking adaptability ladder test (WALT) is a novel test for measuring stepping precision. A standardised ladder is placed on the floor. It consists of 19 rectangular planes which gradually decrease two centimetres in length (range: 64cm - 28cm). Patients starts in the biggest plane and walk as fast as possible to the other side, turn and return to the biggest plane whilst avoiding the ladder rungs. Scoring is via a time score: faster is indicative of better stepping precision. Patients perform the test four times: Twice with one feet per plane, and twice with both feet in one plane.
Mean changes in spatio-temporal gait parameters | Pre C-mill intervention (experimental group week 0, control group week 6), post C-Mill intervention (experimental group week 6, control group week 12) and after the follow-up period of fifteen weeks (experimental group week 21, control group week 27)
  Gait analysis is performed at the movement lab (Radboudumc, Nijmegen). Spatio-temporal parameters are assessed during a 3D full body gait analysis using the VICON analysis system ((©Vicon Motion Systems Ltd., London, UK). Eight infrared cameras measured the coordinates of the reflective markers. The following temporal gait parameters are assessed: stride length (m), step length (m), step width (m), duration of swing time (%), stance time (%), single support (%) and double support (%). Participants walk at their self-selected and maximum speed over a 10 meter walkway.

CONTACTS AND LOCATIONS:
Overall Officials: A.C.H. Geurts, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud universitair medisch centrum, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nonnekes J, van Lith B, van de Warrenburg BP, Weerdesteyn V, Geurts ACH. Pathophysiology, diagnostic work-up and management of balance impairments and falls in patients with hereditary spastic paraplegia. J Rehabil Med. 2017 May 16;49(5):369-377. doi: 10.2340/16501977-2227. PMID 28471471
- [Background] Heeren A, van Ooijen M, Geurts AC, Day BL, Janssen TW, Beek PJ, Roerdink M, Weerdesteyn V. Step by step: a proof of concept study of C-Mill gait adaptability training in the chronic phase after stroke. J Rehabil Med. 2013 Jul;45(7):616-22. doi: 10.2340/16501977-1180. PMID 23811818
- [Background] Fonteyn EM, Heeren A, Engels JJ, Boer JJ, van de Warrenburg BP, Weerdesteyn V. Gait adaptability training improves obstacle avoidance and dynamic stability in patients with cerebellar degeneration. Gait Posture. 2014;40(1):247-51. doi: 10.1016/j.gaitpost.2014.04.190. Epub 2014 Apr 24. PMID 24786476
- [Background] Salinas S, Proukakis C, Crosby A, Warner TT. Hereditary spastic paraplegia: clinical features and pathogenetic mechanisms. Lancet Neurol. 2008 Dec;7(12):1127-38. doi: 10.1016/S1474-4422(08)70258-8. PMID 19007737
- [Derived] van de Venis L, van de Warrenburg BPC, Weerdesteyn V, van Lith BJH, Geurts ACH, Nonnekes J. Improving gait adaptability in patients with hereditary spastic paraplegia (Move-HSP): study protocol for a randomized controlled trial. Trials. 2021 Jan 7;22(1):32. doi: 10.1186/s13063-020-04932-9. PMID 33413555